CLINICAL TRIAL: NCT07010705
Title: Digital Measures for Clinical Trial Endpoints in Huntington's Disease (MEND-HD)
Brief Title: Digital Measures for Clinical Trial Endpoints in Huntington's Disease
Acronym: MEND-HD
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamie Adams, Associate Professor - Department of Neurology, University of Rochester
Other Study IDs: STUDY00010159; 1U01FD008429-01 (FDA)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Huntington Disease; Healthy
Keywords: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- 20 HD-ISS Stage 2: (CAG ≥ 40 and sign/symptom of HD) with or without a support person or family member
  Interventions: Device: ActiGraph LEAP; Device: Axivity AX6
- 20 HD-ISS mild or moderate Stage 3: (CAG ≥40 and sign symptom and functional impact) with or without a support person or family member
  Interventions: Device: ActiGraph LEAP; Device: Axivity AX6
- 20 Healthy controls: age and sex-matched
  Interventions: Device: ActiGraph LEAP; Device: Axivity AX6

INTERVENTIONS:
Device: ActiGraph LEAP — The ActiGraph LEAP has received 510(k) clearance from the US FDA and offers extensive sensor collections, providing continuous digital measures of activity, sleep, mobility, and additional vital signs, including heart rate and variability, oxygen saturation, and skin temperature, in a single fit-for-purpose device.
Device: Axivity AX6 — The Axivity AX6 is a data logger capable of recording raw data from a suite of integrated sensors. It features a state of the art 6-Axis movement sensor measuring linear acceleration and angular velocity at high precision. All sensor locations and Orientations are identical to the AX3 for maximum compatibility. All data is stored in its raw, unaltered format on the embedded flash memory.

SUMMARY:
MEND-HD is a longitudinal study evaluating the feasibility of passive monitoring of gait and chorea in patients with HD and the meaningfulness of these outcomes for patients with HD and their care partners/support persons.

Participants will take part in four virtual visits with study investigators to answer survey questions on movement and cognition, perform in-home movement assessments, and take part in an interview regarding the meaningfulness of gait and chorea in their daily lives.

Participant and care partner interviews will be used for symptom mapping and qualitative data analysis to assess the relevance and impact of the targeted symptoms on the participant's daily life.

The study may be extended to 3 years to include yearly visits.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for participants with adult-onset HD:

* Age of 25-65 years.
* Genetically confirmed HD with CAG >= 40 (HD-ISS Stage 2 or mild/moderate Stage 3)
* English speaking.

Inclusion Criteria for control participants:

* Age of 25-65 years.
* English speaking.

Inclusion Criteria for support persons:

* Self-identified support person or family member of the enrolled participants with HD.
* 18 years or older
* English speaking.

Exclusion Criteria:

* Diagnosis of juvenile-onset HD.
* History of co-morbid neurological disease or disorders such as stroke, multiple sclerosis, or moderate to severe
* Traumatic Brain Injury.
* Use of an assistive device for ambulation.
* Montreal Cognitive Assessment (MoCA) score of 18 or lower
* Acute or chronic medical conditions that significantly impact gait or mobility in the opinion of the investigator, e.g. ankle sprain or fracture, or any orthopedic,
* cardiovascular or psychiatric disease.
* Pregnancy
* Cannot be enrolled into a blinded intervention trial at Baseline

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll 60 participants: 20 HD-ISS Stage 2 (CAG ≥ 40 and sign/symptom of HD) with or without a support person or family member; 20 HD-ISS mild or moderate Stage 3 (CAG ≥ 40 and sign symptom and functional impact) with or without a support person or family member; and 20 controls (age and sex-matched). Participants will not be excluded based on ethnicity, and no subpopulations will be excluded from this study. We will exert specific efforts to ensure the inclusion of minorities, including the Black and Hispanic populations
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Inter-Method Reliability of Total Time in Chorea (Trunk-Worn vs. Wrist-Worn Device) | 1 week
  Total time in chorea is calculated by summing the duration of all bouts of detected chorea throughout each day and then summed across the week (normalized to wear time). The outcome will assess the ability of the wrist-worn device to differentiate between HD and control participants.
Known Group Validity of Total Time in Chorea (Trunk-Worn Device) | 1 week
  Total time in chorea is calculated by summing the duration of all bouts of detected chorea throughout each day and then summed across the week (normalized to wear time). The outcome will assess the ability of the wrist-worn device to differentiate between HD and control participants.
Known Group Validity of Total Time in Chorea (Wrist-Worn Device) | 2 weeks
  Total time in chorea is calculated by summing the duration of all bouts of detected chorea throughout each day and then summed across the week (normalized to wear time). The outcome will assess the ability of the wrist-worn device to differentiate between HD and control participants.
Inter-Method Reliability of Stride Time Variability (Trunk-Worn vs. Wrist-Worn Device) | 1 week
  Stride time variability is defined as the coefficient of variation of stride time, with the median value calculated across all walking bouts lasting at least 10 seconds. The outcome will assess the agreement between trunk-worn and wrist-worn devices among HD and control participants.
Known Group Validity of Stride Time Variability (Trunk-Worn Device) | 1 week
  Stride time variability is defined as the coefficient of variation of stride time, with the median value calculated across all walking bouts lasting at least 10 seconds. The outcome will assess the ability of the trunk-worn device to differentiate between HD and control participants.
Known Group Validity of Stride Time Variability (Wrist-Worn Device) | 2 weeks
  Stride time variability is defined as the coefficient of variation of stride time, with the median value calculated across all walking bouts lasting at least 10 seconds. The outcome will assess the ability of the wrist-worn device to differentiate between HD and control participants.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided